CLINICAL TRIAL: NCT00846508
Title: Phase III Randomized Trial of Comparing CCRT vs. RT Alone for Cervical Cancer Patients Primarily Treated by Radiotherapy and With Clinically Defined Good-prognosis
Brief Title: Cisplatin Based Chemoradiation v.s Radiotherapy for Cervical Cancer and With Clinically Defined Good Prognosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Department of Obstetrics & Gynecology, Chang Gung Memorial Hospital,LIN KOU
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 97-1166A3
Record Dates: First submitted 2009-02-11; First posted 2009-02-18 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; Cisplatin; chemoradiation
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ciaplantin,cancer,survival (Experimental)
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Cisplatin is available commercially as a sterile lyophilized white power in single-dose amber vials containing 10 mg or 50 mg of cisplatin for administration by IV infusion. Every effort should be made to obtain and record the lot numbers of the batches of cisplatin used. Unopened vials of cisplatin are stable for the shelf-life indicated on the package when stored in accordance with the manufacturers' instructions.
  Other Names: Platinex (Cisplatin)

SUMMARY:
This phase III study is designed to examine if low-risk, as defined by clinical and radiological parameters, stage IB-IIB cervical cancer patients treated by cisplatin-based chemoradiation, which is a recommended method by today's standard, have greater toxicities but similar survival rate as those treated by radiotherapy (RT) alone. Patients will be primarily treated with radiotherapy with same protocol, but without concurrent chemotherapy in the control arm, and with weekly cisplatin (40 mg/M2) for 6 courses in the study arm. This study will be conducted at all branches of Chang Gung Memorial Hospital except Chia-I.

Patients will be randomized to either arm after stratification of risk factors. Each arm will recruit 104 patients who have no LN and systemic metastasis as defined by CT/MRI and FDG-PET. The primary end point is grade 3-5 late toxicities, and secondary end points are 1) recurrence free survival; 2) acute toxicity of treatments; 3) sites of recurrence; 4) quality of life; 5) total treatment time. It is expected to take 5 years to recruit enough case number.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objectives:

•To examine if low-risk, as defined by clinical and radiological parameters, stage IB-IIB cervical cancer patients treated by cisplatin-based CCRT have greater toxicities but similar survival rate as those treated by RT alone.

Secondary Objectives:

•To conduct a translational research to find out the molecular markers associated with radiosensitivity and distant metastasis in cervical cancer patients.

104 cases for each arm.(total 208 cases)

Radiotherapy will start within 3 weeks of randomization.

Chemotherapy:

Cisplatin 40mg/M2 IV infusion weekly concurrently with radiotherapy, up to 6 courses.

Investigation during treatment (for patients on both arms)

1. . Hematology: A complete blood count is required at weekly intervals.
2. . Renal function: Serum creatinine is required before each course of CT.
3. . Body weight and performance status: will be evaluated on the day of weekly visit on radiotherapy clinics. Performance status is graded by ECOG scale.
4. . Quality of life assessment: assess by EORTC-C30 & CX28 scales at pre-RT, 3-4 weeks and 6-7 weeks during RT.

Investigation during follow-up:

When radiotherapy (RT) treatment is completed, patients will be followed up as out-patients basis. The first visit will be within 2 months after last RT. For patients whose tumor does not regress completely at the end of RT, monthly follow-up for at least 3 months or to the time of complete regression is recommended. After first follow-up or time of compete regression of tumor, patients will be followed up at 3-monthly intervals for 2 years, 4-monthly for one year, then 6-monthly.

Quality of life assessment: assess by EORTC-C30 & CX28 scales at 2 months, 4-5 months after RT, then q 6 months x 2 and yearly for another 2 years.

Dosage modification and toxicity Toxicity must be recorded at each attendance for chemotherapy and monthly during radiotherapy on the "on study form".

1. . Hematological toxicity: ANC < 1500 /mm3 and/or platelet < 100,000 /mm3 prior to chemotherapy will require one week delay in treatment until these levels have been reached. If the parameters are still below requirements 1 week later, administration of chemotherapy could still be proceeded if 1000 <ANC < 1500 /mm3, platelet > 50,000 /mm3 at reduced dose (25% off).

   Radiotherapy will not be delayed unless severe infection or a white count less than 1000/mm3
2. . Renal toxicity:

   a). Cisplatin: Serum creatinine < 1.5 mg% (creatinine clearance > 70 ml/min): full dose; 1.6-1.9 mg% (or 0.6-0.8 mg% above base line, or Ccr 50-70 ml/min): 25% off; > 2.0 mg% (or > 1.2 mg% over baseline or 50% decrease of Ccr): no cisplatin
3. . Neurotoxicity: Cisplatin discontinued on Grade 3 neuropathy. 30% dose decrease for Grade 2 neurotoxicity or ototoxicity
4. . Ototoxicity: Ototoxicity is rare within 4 -6 courses or cisplatin, but if clinical significant deterioration of hearing loss (grade 3) was noted, cisplatin will be discontinued. The aged are more susceptible to ototoxicity.
5. . Genitourinary complications Urinary tract infection or radiation cystitis may be noted during the course of treatment, CT or CT+RT will be withheld in case of grade 3 toxicity
6. Gastroenterological toxicity:

Acute radiation enteritis may prelude continuation or delay either CT or CT+RT

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed squamous cell carcinoma of cervix
* Clinical FIGO stage IB-IIB
* Planned to be primarily treated by RT.
* Age: 45 < age< 80
* No enlarged pelvic or para-aortic LN shown in CT-MRI (by CT-MRI criteria) and positive LN in FDG-PET studies.
* Patients must have adequate bone marrow, pulmonary, liver and renal function
* The interval between RT and randomization is not greater than 6 weeks.
* Performance status
* Patients must have signed informed consent to participate this study

Exclusion Criteria:

* Age ≧80 or <=45
* Documented pelvic LN or extrapelvic metastases: para-aortic LN, lung, liver
* LN-positive on PET scans.
* General medical condition or attitude makes them unsuitable for cisplatin therapy.
* Small cell carcinoma, adenocarcinoma or adeno-adenosquamous carcinoma.
* Previous pre-RT chemotherapy or pelvic RT

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
As defined by clinical and radiological parameters, stage IB- IIB cervical cancer patients treated by cisplatin-based CCRT have greater toxicities but similar survival rate as those treated by RT alone | 2012

SECONDARY OUTCOMES:
To conduct a translational research to find out the molecular markers associated with radiosensitivity and distant metastasis in cervical cancer patients. | 2013

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Hong Hong, M.D, Principal Investigator — Department of Radiation Oncology,LIN KOU
Locations (2):
- Taiwan (2):
  - Chang Gung Memory Hpspital, Kaohsiung City
  - Chang Gung Memory Hpspital, Keelung